CLINICAL TRIAL: NCT03657030
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Study of Escalating Single and Multiple Doses of CVN424 in Healthy Subjects
Brief Title: Study of CVN424 in Healthy Subjects
Acronym: CVN424
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevance Beta, Inc. (Industry)
Responsible Party: Sponsor
Organization: CerevanceBeta (Unknown)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: CVN424-101
Record Dates: First submitted 2018-08-24; First posted 2018-09-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Single ascending dose and multiple ascending dose study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Active Comparator): The planned dose levels will be 1, 5, 25, 75, and 225 mg CVN424 and matching placebo.
  Interventions: Drug: CVN424; Drug: Placebo
- Multiple Ascending Dose (Active Comparator): The planned dose levels will be 25, 75, and 150 mg CVN424 and matching placebo.
  Interventions: Drug: CVN424; Drug: Placebo

INTERVENTIONS:
Drug: CVN424 — SAD / MAD
Drug: Placebo — Placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, single- and multiple-dose ascending study in healthy subjects.

DETAILED DESCRIPTION:
Part 1: Single-Dose Regimen and Fasted-Fed Crossover - For the single-dose regimen, approximately 40 healthy male and female subjects will be enrolled in 1 of 5 single dose cohorts (designated as S1 through S5, respectively) in an ascending fashion.

Part 2: Multiple-Dose Regimen

- For the multiple-dose regimen, approximately 24 healthy male and female subjects age 18 to 50 years old will be enrolled in 1 of the 3 multiple-dose cohorts (designated as M1 through M3, respectively) in an ascending fashion.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Investigator, the subject is capable of understanding and complying with protocol requirements.
* The subject signs and dates a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures.
* Subject is a healthy male or female adult who is 18 to 50 years of age inclusive at the time of ICF and study drug dosing.
* Subject weighs at least 45 kg (99 lbs) and has a BMI between 18.0 and 30.0 kg/m2, inclusive at Screening.
* A male subject who is nonsterilized and sexually active with a female partner of childbearing potential* agrees to use adequate contraception* from signing of the ICF throughout the duration of the study and for 12 weeks after last dose.
* A female subject with no childbearing potential, defined as the subject has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (defined as continuous amenorrhea of at least 2 years and FSH>40 IU/L).

Exclusion Criteria:

* Subjects have a known hypersensitivity to any component of the formulation of CVN424.
* Subjects have evidence of CS neurologic, cardiovascular, pulmonary, hepatic, hematopoietic disease, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, serious allergy, allergic skin rash, psychiatric disorder, or other abnormality that may impact the ability of the subject to participate or potentially confound the study results.
* There is any finding in the subject's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a condition that might interfere with the conduct or interpretation of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events | Baseline through 14 days post-dose
  Occurrence of all adverse events from signing of informed consent through end of study treatment.
Evaluation of Hematology | Baseline through 14 days post-dose
  RBC
Evaluation of Vital Signs | Baseline through 14 days post-dose
  Oral Temperature (°C )
Evaluation of Electrocardiograms | Baseline through 14 days post-dose
  Standard 12-lead ECG - QT interval
Evaluation of BMI | Baseline through 14 days post-dose
  Weight and Height will be combined to calculate BMI using the following formula: BMI = weight (kg)/[height (m)]2
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  ALT
Evaluation of Urinalysis | Baseline through 14 days post-dose
  pH
Evaluation of Vital Signs | Baseline through 14 days post-dose
  Respiration rate
Evaluation of Vital Signs | Baseline through 14 days post-dose
  Pulse rate
Evaluation of Vital Signs | Baseline through 14 days post-dose
  Blood pressure (both systolic and diastolic)
Evaluation of Hematology | Baseline through 14 days post-dose
  WBC with differential (%and absolute) platelets, PT/INR
Evaluation of Hematology | Baseline through 14 days post-dose
  Hemoglobin
Evaluation of Hematology | Baseline through 14 days post-dose
  Hematocrit
Evaluation of Hematology | Baseline through 14 days post-dose
  PT/INR
Evaluation of Hematology | Baseline through 14 days post-dose
  Platelets
Evaluation of Electrocardiograms | Baseline through 14 days post-dose
  Standard 12-lead ECG- QTcB interval
Evaluation of Electrocardiograms | Baseline through 14 days post-dose
  Standard 12-lead ECG - QTcF interval
Evaluation of Electrocardiograms | Baseline through 14 days post-dose
  Standard 12-lead ECG - RR interval
Evaluation of Electrocardiograms | Baseline through 14 days post-dose
  Standard 12-lead ECG - QRS interval
Evaluation of Electrocardiograms | Baseline through 14 days post-dose
  Standard 12-lead ECG - PR interval
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Albumin
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Alkaline phosphatase
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Lipase
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  AST
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Total bilirubin
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Direct bilirubin
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Total protein
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Creatinine
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Blood urea nitrogen
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Creatine kinase Glucose, Chloride, Bicarbonate
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  GGT
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Potassium
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Sodium
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Glucose
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Chloride
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Bicarbonate
Evaluation of Serum Chemistry | Baseline through 14 days post-dose
  Calcium
Evaluation of Urinalysis | Baseline through 14 days post-dose
  Specific gravity
Evaluation of Urinalysis | Baseline through 14 days post-dose
  Protein
Evaluation of Urinalysis | Baseline through 14 days post-dose
  Glucose
Evaluation of Urinalysis | Baseline through 14 days post-dose
  Blood
Evaluation of Urinalysis | Baseline through 14 days post-dose
  Nitrite
Evaluation of Urinalysis | Baseline through 14 days post-dose
  Microscopic Analysis (only if positive dipstick results): RBC/high power field, WBC/high power field, Epithelial cells, casts

SECONDARY OUTCOMES:
Plasma Concentration (AUC) of CVN424 | SAD: PK Collection on Day 1-4, and early termination (up to 8 days); MAD: PK Collection on Day 1-10, and early termination (up to 14 days)
  To evaluate the pharmacokinetics of single and multiple doses of CVN424. Pharmacokinetic parameters including, but not limited to area under the plasma concentration-time curve (AUC) from 0 to 24hours (AUC0-24)
Plasma Concentration (Cmax) of CVN424 | SAD: PK Collection on Day 1-4, and early termination (up to 8 days); MAD: PK Collection on Day 1-10, and early termination (up to 14 days)
  To evaluate the pharmacokinetics of single and multiple doses of CVN424. Pharmacokinetic parameters including, but not limited to maximum plasma concentration (Cmax).
Food effect by measurement of plasma PK (Cmax) | Baseline through 14 days post-dose
  Assess the effect of food on the bioavailability in the current formulation after digesting a high caloric meal.
Food effect by measurement of plasma PK (AUC) | Baseline through 14 days post-dose
  Assess the effect of food on the bioavailability in the current formulation after digesting a high caloric meal.

OTHER OUTCOMES:
DNA isolation and genotyping | Day 1
  Drug metabolic enzyme and transporter polymorphisms that may contribute to variability in CVN424 will be reported.
  Single-dose -pre-dose
  Multi-dose
  -pre-dose
RNA isolation and genotyping | Day 1 and Day 7
  Single-dose -pre-dose, 8 and 24 hours post dose
  Multi-dose
  -pre-dose, 8 and 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: David H Margolin, MD, PhD, Study Director — Cerevance, Inc.
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No